CLINICAL TRIAL: NCT01211067
Title: Histological Findings of the Internal Inguinal Ring in Patients With Indirect Inguinal Hernia
Brief Title: Study of Histological Findings of the Internal Inguinal Ring in Patients With Indirect Inguinal Hernia
Status: Completed | Type: Observational
Sponsor: Cirujanos la Serena (Other)
Responsible Party: Marcelo A. Beltrán, Hospital de La Serena
Other Study IDs: HLS-0015-1109
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Last update posted 2010-09-29 (Estimated); Status verified 2010-09

CONDITIONS: Indirect Inguinal Hernia
Keywords: Inguinal hernia; Inguinal ring; Histology; Hernioplasty; Lichtenstein
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A 1 cm tissue sample of the internal inguinal ring taken during elective hernioplasty
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients age: 15 - 40 years-old: Patients within the 15 to 40 years-old age-group
  Interventions: Procedure: Lichtenstein hernioplasty
- Patients age: 41 to 60 years-old: Patients within the group-age from 41 to 60 years-old
  Interventions: Procedure: Lichtenstein hernioplasty
- Patients age: older than 61 years-old: Patients within the group-age from 61 years-old and older
  Interventions: Procedure: Lichtenstein hernioplasty

INTERVENTIONS:
Procedure: Lichtenstein hernioplasty — * Mesh hernioplasty
  * Ultrapro mesh (Ethicon, Johnson & Johnson)

SUMMARY:
The histology of the internal inguinal ring in patients with indirect hernia submitted to elective surgery was studied. In contrast with recently published studies, the investigators believe that histological findings of the internal inguinal ring would reflect those associated and expected with normal aging.

ELIGIBILITY:
Inclusion Criteria:

* Male gender
* Older than 15 years-of-age
* Unilateral indirect inguinal hernia
* Non-smokers
* Non-diabetics
* Non-connective tissue conditions
* Primary inguinal hernia

Exclusion Criteria:

* Female gender
* Younger than 15 years-of-age
* Bilateral inguinal hernia
* Direct or combined direct-indirect inguinal hernia
* Femoral hernia
* Smokers
* Diabetics
* Other connective tissue diseases
* Recurrent inguinal hernia

Min Age: 15 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with indirect inguinal hernia submitted to elective surgery with the Lichtenstein hernioplasty technique
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2009-09; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Histology of the internal inguinal ring | 6 months
  Histology and histological findings of the internal inguinal ring in patients submitted to elective surgical reparation of an indirect inguinal hernia

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo A Beltrán, M.D., Principal Investigator — Hospital de La Serena
Locations (1):
- Hospital de La Serena, La Serena, Coquimbo Region, Chile

REFERENCES:
- [Background] Barria C, Beltran MA, Contreras MA, Cruces KS. Histology of the internal inguinal ring: it is really a novelty? Hernia. 2010 Jun;14(3):339-40. doi: 10.1007/s10029-010-0661-4. Epub 2010 May 1. No abstract available. PMID 20437189